CLINICAL TRIAL: NCT01668030
Title: Comparison of Wound Bed Establishment in Facial Burns Using Two Standard Ointments
Brief Title: Comparison of Wound Bed Establishment in Facial Burns
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 11.0456
Record Dates: First submitted 2012-08-08; First posted 2012-08-17 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Burns
Keywords: Facial; Partial thickness
MeSH Terms: conditions — Burns; Facies | interventions — Bacitracin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants received both the test drug and the standard of care, one on each side of the face.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bacitracin on left, Enzymatic agent on right (Experimental): Subjects were randomized to receive enzymatic agent on right side of face and bacitracin on left.
  Interventions: Drug: Enzymatic agent; Drug: Bacitracin
- Bacitractin on right, enzymatic agent on left (Experimental): Subjects were randomized to receive enzymatic agent on left side of face and bacitracin on right.
  Interventions: Drug: Enzymatic agent; Drug: Bacitracin

INTERVENTIONS:
Drug: Enzymatic agent — Enzymatic agent
Drug: Bacitracin

SUMMARY:
Forty percent of patients admitted to the contributing regional burn unit over a five month period received facial burns (n=14). The purpose of this study is to examine if the time until a granulation bed is well established can be decreased be using an enzymatic agent, when compared to a second standard ointment, for patients with partial-thickness facial burns. The current study will use a prospective, experimental study design in which each individual will be their own matched control. That is, each individual will receive both the experimental ointment (one-side of the face) and the standard ointment (other-side of the face). Outcomes measured will be the benefits (e.g., decreased in the time until granulation bed establishment) one ointment achieves in partial-thickness facial burns when compared to a second ointment. Exploratory analyses will examine the relationships among demographic variables, granulation bed establishment time, pain, anxiety, itching, and scarring. That is, testing whether the time until granulation establishment may be associated with an individual's demographic variables, treatment type, pain, anxiety, itching levels, and scarring. Significance for all analysis will be at the 0.05 level. The investigators hypothesize that promoting rapid granulation bed establishment will decrease hospital length of stays, costs, risk of infection, and possibly associated appearance changes. The results from the current study will provide preliminary findings for a future, more sophisticated study.

DETAILED DESCRIPTION:
Rapid wound healing in burn injuries advances wound closure, and decreases opportunities for infection and scarring (Hansbrough, Achauer, Dawson, et al., 1995; Soroff & Sasvary, 1994); also leading to a shorter length of stays (LOS). Decreased LOS in the hospital supported by rapid wound closure facilitates reentry to the home and work environments should lead to a reduction in the costs associated with hospitalization. In addition, for patients with facial burns, rapid granulation bed establishment may decrease associated appearance changes.

Use of an enzymatic agent has been described in only three studies (Hansbrough, Achauer, Dawson, et al., 1995; Soroff & Sasvary, 1994; Varma, Bugatch, & German 1973). Treatment an enzymatic agent resulted in shorter time to achieve a clean wound bed and significantly more rapid wound healing when compared to controls or other agents for 94 patients with non-facial, partial-thickness burns (Hansbrough, Achauer, Dawson, et al.; Soroff & Sasvary). Twenty patients with dermal ulcers treated with an enzmatic agent, when compared to placebo controls, showed significantly decreased pus, odor, necrosis, and inflammation (Varma, Bugatch, & German, 1973). There was a relative reduction in wound size almost reaching significance (p<0.07) for those patients with dermal ulcers too.

Though an enzymatic agent is without purported antibiotic properties, a rapid reduction in bacterial burden in wounds has been shown in animal models (Payne, Salas, Ko, Naidu, Donate, Wright et al., 2008). The bacterial burden decreased rapidly in scald burn wounds to achieve a bacterial balance for 15 rats with E-coli infected wounds when compared with saline-treated controls to <105 colony forming units/gram of tissue (p < .05).

Previous studies have suggested that the exploratory variables being collected are associated with shorter healing times and lower infection rates. Whether these differences are actually due to some other mediating/moderating factor (gender-specific enzyme or hormone concentrations, gene interaction, metabolism, etc) and not the exploratory variables is unclear and not empirically established. A future, larger study will hopefully more fully explore these relationships. However, to justify the more detailed investigations will require showing differences at the more crude level. Unfortunately, to date there has been no research examining the potential benefits of using collagenase in patients with facial burn injuries. As a result, the aims of this study are to:

1. Show the benefit (e.g., decreased time until the granulation bed is well established, shorter time until wound closure) an enzymatic agent achieves in partial-thickness facial burns when compared to a common antibacterial agent;
2. Investigate the interrelationships among demographic variables, treatment, pain, anxiety, and itch;
3. Explore whether time to granulation bed establishment can be predicted from treatment; when adjusting for demographic variables, pain, anxiety, and itch levels.
4. Examine the long-term scarring and social experience of persons with facial burns.

Design: A prospective, experimental study design in which each individual will be their own matched control.

Methods

Procedure. Within 24 hours of burn unit admission, patients or their spouses, or guardians will be asked regarding study participation. Upon patient agreement, and signing the institutional review board approved informed consent form, HIPAA Research Authorization, a demographic information form will be completed and wound culture results obtained (if ordered).

The patients will be randomized into receiving either bacitracin or collagenase to the right side of the face (ointment one). Ointment two will be applied to the left side of the face. Treatment of the partial-thickness facial burns will be performed by the nurses on the burn unit according to burn unit protocol. Therefore, each person will serve as their own matched control, thus reducing the sample size required to achieve sufficient power for the study by reducing deviance between cases and control (i.e., age, pain, itch, size of burn, and scarring). Also, this type of study design will allow us to achieve valid, reliable results with fewer individuals. This is a typical study design for similar ointment and eye drops studies. The bridge of the nose will be used as a guide to divide the face in half lengthwise. The wound will be cleansed and dressed twice daily. Treatment will continue until the granulation bed is well established. Daily ratings of pain, anxiety, and itch will be obtained at each morning dressing change. Digital photographs of only the facial burn will be taken weekly and at the first outpatient visit.

Patient confidentiality will be maintained by assigning participants a random, unique, study identification number that cannot be linked directly to any individual. This random number will be used in all study data sets for data management and data analysis. Signed (approved) informed consent forms will be kept in a locked file in the principle investigator's office. The research data sets will be stored on a university secured computer drive.

Digital photographs will be identified by patient number. These photographs will be rated by burn wound experts recruited from a posting on the American Burn Association web site (e.g. nurses and/or physical therapists certified in wound care with a minimum of 5 years' experience). Patients' records will also be assessed weekly as to whether any patient on study has a wound or blood infection confirmed by a positive laboratory culture. Those patients with confirmed positive cultures will be dropped from the study. Patient pain, anxiety, and itch scoring will be obtained and recorded by the nurses caring for patients on the burn unit.

Assessment of scarring will be obtained at the first out-patient visit by both the healthcare provider and patient. For the three and six month follow-ups, every effort will be made to have both the health care provider and patient assessments, however, it may not always be possible to have the patient return to the hospital (e.g., costs associated with travel and missing work) so the patient's assessment will be obtained via telephone. Assessment of the social experience will be obtained by completing the two instruments and open-ended questions either in-person or through a telephone interview at the first out-patient visit, at three and six months after injury.

Instrumentation

Pain and Anxiety. Physician ordered analgesic and anxiety therapy will be provided per patient request prior to each dressing change. At each morning dressing change, patients will rate their perception of pain and anxiety, separately, with a 10-point visual analogue scale (where 1= no pain, or anxiety and 10= the most possible) at three time points. These times will be: prior to cleansing and debridement, at completion of the dressing change, and 30 minutes after treatment. The Richmond Agitation and Sedation Scale (RASS) will be used with non-verbal patients.

Richmond Agitation and Sedation Scale (RASS). Inter-rater reliability in 290-paired observations by nurses, results of both the RASS demonstrated excellent inter-rater reliability (weighted kappa, 0.91 and 0.94, respectively) (Ely, Truman, Shintani, et al., 2003). Criterion validity was tested in 411-paired observations in the first 96 patients of the validation cohort, in whom the RAS showed significant differences between levels of consciousness (P<.001 for all) and correctly identified fluctuations within patients over time (P<.001). Face validity was demonstrated via a survey of 26 critical care nurses, which the results showed that 92% agreed or strongly agreed with the RASS scoring scheme, and 81% agreed or strongly agreed that the instrument provided a consensus for goal-directed delivery of medications.

Itch. Physician ordered itch therapy (e.g., Benadryl, Atarax, or Claritin) will be provided per patient request prior to each dressing change. At each morning dressing change, patients will rate their perception of itch with a 10-point visual analogue scale (where 1=no itch and 10=the most possible), at three time points. These times will be: prior to cleansing and debridement, at completion of the dressing change, and 30 minutes after treatment.

Scarring. Scarring will be measured by two instruments [The Patient and Observer Scar Assessment Scale (POSAS)] developed by Draaijers, Tempelman, Botman, et al. (2004) and further tested by Van de kar, Corion, Smeulders, et al. (2005. These two instruments, one for the health care provider and the second for the patient, recognizes the need for both the professional's and patient-based need for scar assessment, whereas, the Vancouver Scar Scale (VSS) only assesses scar severity from the professional's viewpoint. Though the VSS has been accepted and used as a scar assessment tool, there is not evidence to suggest it is the "gold standard" measure of burns scarring, and additionally, it does not include the patient's perception of their scarring.

The POSAS has items assessing vascularity, pigmentation, thickness, relief and pliability, rated on a 10-point numeric scale, with normal skin and worst scar used as end labels. Items on the patient scale directly correspond to theses except for scar color. Patients are asked to rate their itchiness and scar pain. A ten-point numeric scale is used (1=no complaints /normal skin, 10=worst imaginable/very different). Individual items are summed with higher scores representing poorer scars and lower scores representing scars more closely to normal skin. Both scales showed acceptable internal consistency (Cronbach's alpha 0.76 (patient) and 0.69 (observer). The test-retest reliability of the patient scale has not been evaluated in burn scars.

Social Experience. It is proposed that partial-thickness burns to both sides of the face result in non-normal appearance which may cause stigmatizing and dehumanizing behavior directed at these burn survivors (Lawrence, Fauerbach, Heinberg, Doctor, and Thombs, 2006; Lawrence, Rosenberg, Rimmer, Tombs, and Fauerbach, 2010). The following two instruments will assess the social experience.

The social experience will be measured by two instruments: the Perceived Stigmatization Questionnaire (PSQ) and the Social Comfort Questionnaire (SCQ) (Lawrence, Fauerbach, Heinberg, Doctor, and Thombs, 2006; Lawrence, Rosenberg, Rimmer, Tombs, and Fauerbach, 2010). Both instruments were developed and tested for use with a population of burn injury survivors. The PQS is a 21 item scale where each item is measured on a 5-point Likert scale (never, almost never, sometimes, often, always). Three factors were loaded: absence of friendly behavior, confused behavior and starring, and hostile behavior. Scores are calculated by totaling items and dividing by 21. Higher scores indicate levels of perceived stigmatizing behaviors.

The SCQ is an eight item, one factor scale. Each item is also measured on a 5-point Likert scale (never, almost never, sometimes, often, always). The final score is the average of items; higher scores indicate higher social comfort.

Open-ended Questions: Several open-ended questions will be included to allow participants to describe instances of how their social experience changed after the facial burn injury. It is hoped that these answers will further clarify the two instrument findings

ELIGIBILITY:
Inclusion Criteria:

* patients (over the age of 18 years) admitted to the burn unit with a minimum of 1% partial-thickness burns each side of the face.

Exclusion Criteria:

* patients with superficial or full-thickness facial burns;
* patients receiving facial grafts; patients with burns from chemical or contact sources;
* patients with wound infection;
* any patients starting treatment 24 hours after burn injury;
* patients with known sensitivity to either standard treatment; and
* any women by history who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlee R. Lehna, PhD, APRN-BC, Principal Investigator — University of Louisville, School of Nursing
Locations (1):
- UofL Health Care, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from hospital burn unit.
Units Other Than Participants: Cheek (side of face)
Groups:
- Bacitracin Treated Side of Face: Bacitractin was applied to one side of face.
- Enzymatic Agent Treatment Side of Face: Enzymatic agent applied to cheek
Period: Overall Study
Arm/Group | Bacitracin Treated Side of Face | Enzymatic Agent Treatment Side of Face
Started | 10; 10 Cheek (side of face) | 10; 10 Cheek (side of face)
Completed | 10; 10 Cheek (side of face) | 10; 10 Cheek (side of face)
Not Completed | 0; 0 Cheek (side of face) | 0; 0 Cheek (side of face)

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Double Blind (masked to subject, caregiver, & outcome assessor. Intervention is that either drug is randomized into being applied to either right or left side of face.
  Enzymatic treatment versus Bacitracin: Person is their own control. Ointments randomly applied to either side of face.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Time to Wound Epithelialization
Description: Time it required the subjects treated with two standard ointments to establish a wound bed.
Time Frame: Two years
Measure: Number; unit: days
Units Other Than Participants: cheeks (side of face)
Groups:
- Bacitracin Treated Side of Face; Enzymatic Agent Treatment Side of Face: Double Blind (masked to subject, caregiver, & outcome assessor. Intervention is that either drug is randomized into being applied to either right or left side of face.
  Enzymatic agent versus Bacitracin: Person is their own control. Ointments randomly applied to either side of face.
Arm/Group | Bacitracin Treated Side of Face | Enzymatic Agent Treatment Side of Face
Number analyzed (Participants) | 10 | 10
Number analyzed (cheeks (side of face)) | 10 | 10
days | 37.4 | 37.6
Statistical Analysis 1: Comparison: Bacitracin Treated Side of Face vs Enzymatic Agent Treatment Side of Face; Test type: Superiority; p = .0853, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Small sample size. The study did not differentiate between deep partial thickness and superficial partial thickness burns. another way to trial this study methodology would be to use animal subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No